CLINICAL TRIAL: NCT05346549
Title: Energy Regulation and Nutritional Status of Children: A Satiation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ghana (Other)
Collaborators: University of Glasgow (Other); University of Stirling (Other)
Responsible Party: Principal Investigator, Eunice Nortey, Principal Investigator, University of Ghana
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GHS-ERC:022/11/21
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Underweight; Stunting; Healthy
MeSH Terms: conditions — Thinness; Growth Disorders

STUDY DESIGN:
Intervention Model Description: cross-over energy compensation study, participants acting as their own controls
Who Masked: Participant, Investigator
Masking Description: Two similar tasting drinks will be used in random order, one low and one high energy after a standardized meal. The weight of food consumed will be measured by an observer blind to which supplement has been used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High energy (Experimental): Child will be given a high energy drink: sugar free ribena squash (2kcal/100ml) plus a weighed amount of super soluble maxijul. Super Soluble Maxijul is a powdered carbohydrate energy source, which can be mixed with sweet or savoury foods/ liquids. It is safe for use in both children and adults that require fortification with a high or readily available carbohydrate. It is flavourless and tasteless offering little to no change in taste, flavor and texture of food being added to. It supplies 380 kcal energy per 100g powder. The amount given will supply 10% of the child's daily energy requirements per Kg - for example a 3-year old child weighing about 16 kg requires approximately 1300 kcal/day. Hence the high energy drink will supply the child with 130kcal.
  They will be given 10 minutes to drink the preload and 30 minutes after this they will eat standardized weighed buffet lunch of known energy content suitable for their age, chosen in consultation with the parents.
  Interventions: Behavioral: High energy preload
- Low energy (Experimental): Child will be given a low energy drink of the same volume selected to be as similar as possible to the high energy drink: sugar free ribena squash containing 2kcal per 100ml.
  They will be given 10 minutes to drink the preload and 30 minutes after this they will eat lunch containing the same range of weighed buffet foods as above.
  Interventions: Behavioral: Low energy preload

INTERVENTIONS:
Behavioral: High energy preload — Tests the extent to which participants reduce their food intake at a meal following ingestion of a high energy preload drink.
  Other Names: Satiation study
  Arms: High energy
Behavioral: Low energy preload — Tests the amount participants eat at a meal following ingestion of a low energy preload drink
  Other Names: Satiation study
  Arms: Low energy

SUMMARY:
This is study among children attending child welfare clinics in Greater Accra Region of Ghana. The investigators want to find out if moderately malnourished children regulate the food energy intake similarly to healthy children, using an established method to assess energy compensation.

DETAILED DESCRIPTION:
Malnutrition originates from a complex interplay between genes and environment, manifesting in changes to hormones, metabolism, and behaviour. Energy regulation which determines food intake or avoidance plays a significant role in the cause, prevention and treatment of malnutrition. There is however limited knowledge of how energy regulation develops in children and its effect on their nutritional status in the context of undernutrition in children. A good understanding of energy regulation in children is therefore essential in designing interventions for tackling infant malnutrition.

A standardised energy compensation study will be undertaken in 60 children- 20 moderately malnourished, 20 stunted and 20 healthy. At two visits at least a week apart, the children will be given one of two similar tasting drinks in random order, one with very few calories and another with extra, without them knowing which is which. After 30 minutes they will eat as much as they want of a standardized lunch. All foods and drinks offered will be weighed before and after, to calculate the amount of energy eaten in total after the low energy drink, compared to the high energy drink.

ELIGIBILITY:
Inclusion Criteria:

* moderately malnourished (WHZ between -3 and -2 Z-scores) or stunted (HAZ<-2SD) or Healthy (WHZ >-2SD and HAZ >-2SD) children age 12-36 months.
* Children should be attending child welfare clinics at the selected communities.
* The children should be accompanied by a main caregiver who is actively involved in cooking for and/or feeding the child.
* Children who are able to fast for at least 2 hours prior to the experiment.

Exclusion Criteria:

* Children with congenital disorders, disabilities and diseases requiring specialised care and hospitalisation.
* Children with severe malnutrition with complications that required inpatient care.
* Tube-fed children.
* Children who are both stunted and moderately malnourished

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Compensation index (Compx) | calculated on second visit (1-4 weeks after first visit) after consumption of second test meal
  The difference in energy consumed after high compared to low energy preload as percent of energy in preload. This will be calculated using a mathematical formulae:
  Compx = [ (energy from meal following low energy preload - energy from meal after high energy preload) / (energy from high energy preload - energy from low energy preload) ] x 100%

SECONDARY OUTCOMES:
Difference in total energy consumed | calculated on second visit (1-4 weeks after first visit) after consumption of second test meal
  The total amount of energy consumed from preload plus test meal after high compared to low energy preload

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Nortey, Principal Investigator — University of Ghana
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No
Data may be made available on request